CLINICAL TRIAL: NCT06867471
Title: Effects of Exogenous Ketosis on Proteinuria and Renal Function in Patients with Chronic Kidney Disease and Patients with Polycystic Kidney Disease
Brief Title: Effects of Exogenous Ketosis on Proteinuria and Renal Function
Acronym: KETO-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TZL-2-2024
Record Dates: First submitted 2024-11-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Renal Insufficiency, Chronic; Polycystic Kidney Diseases; Proteinuria; Ketosis
Keywords: Kidney physiology; Glomerular Filtration Rate; Chronic Kidney disease; Ketosis; Proteinuria; Natriuresis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Polycystic Kidney Diseases; Proteinuria; Ketosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ketone-IQ and the placebo drink will be transferred to neutral bottles and relabeled. The local pharmacy will be handling the blinding and randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone diol (Ketone-IQ), then Placebo drink (Other): For four weeks each subject will receive Ketone Diol, R-1,3-butanediol, administered as a drink (Ketone-IQ) twice a day, then crossed over to receive a taste and volume matched placebo drink for four weeks.
  Each individual will receive 400mg/kg before bedtime in addition to 200mg/kg with a minimum of 6 hours in between throughout the treatment period.
  Interventions: Dietary Supplement: Ketone Diol, R-1,3-butanediol (Ketone-IQ); Other: Placebo drink
- Placebo drink, then Ketone diol (Ketone-IQ) (Other): For four weeks each subject will receive a placebo drink twice a day, then crossed over to receive Ketone Diol, R-1,3-butanediol, administered as a drink (Ketone-IQ) twice a day for four weeks.
  Each individual will receive 400mg/kg before bedtime in addition to 200mg/kg with a minimum of 6 hours in between throughout the treatment period.
  Interventions: Dietary Supplement: Ketone Diol, R-1,3-butanediol (Ketone-IQ); Other: Placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone Diol, R-1,3-butanediol (Ketone-IQ) — Effect variables will be measured on the last day of treatment with Ketone-IQ
Other: Placebo drink — Effect variables will be measured on the last day of treatment with Placebo

SUMMARY:
A randomized, placebo-controlled, double-blinded crossover study will be conducted. Fourteen patients with polycystic kidney disease (PKD) and 29 patients with proteinuric kidney disease will receive ketone bodies (Ketone-IQ) and placebo in a randomized order. Each treatment period is four weeks. There will be a wash-out period of two weeks in between treatment periods. Effect variables will be measured in the last day of each treatment period.

DETAILED DESCRIPTION:
Background: Until recently, the only treatment shown to slow progression of chronic kidney disease (CKD) has been angiotensin converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs).

The use of sodium glucose transporter 2 (SGLT2)-inhibitors, which work by blocking the activity of sodium-glucose-cotransporter 2 channels in the proximal kidney tubule, has completely transformed the treatment of proteinuric kidney disease, with a 28% decrease in the risk for cardiorenal outcomes. Despite these new treatment options, a significant proportion of patients still succumb to kidney failure, require hospitalization for heart failure and die prematurely. Thus, additional preventive measures are essential.

Renewed interest in the physiological role of ketone bodies (KB) has emerged. It has become increasingly clear that ketosis has several beneficial effects including anti-epileptic effects, improved exercise capacity, lipid profile, cardiac function and cognition.

However, only few clinical studies have studied renal effects of exogenous ketosis, and to our knowledge there are no clinical studies examining the effects long term effects of renal ketosis in patients with CKD.

Hypothesis: Ketosis decreases urine albumin to creatinine ratio (ACR) and glomerular filtration rate (GFR) in patients with CKD/PKD.

Methods: A randomized, placebo-controlled, double-blinded crossover study will be conducted. Twenty-nine patients with proteinuric kidney disease (study a) and 14 patients with PKD (study b) will receive ketone bodies (Ketone-IQ) and placebo in a randomized order. Each treatment period is four weeks. There will be a wash-out period of two weeks in between treatment periods. Effect variables will be measured in the last day of each treatment period.

Perspectives: The study has the potential to provide information regarding the therapeutic potential of ketone bodies in patients with CKD/PKD.

ELIGIBILITY:
Inclusion Criteria

Study A (patients with CKD):

* ACR > 200 mg/g <3000 mg/g
* eGFR >30 ml/min/1,73m2
* Treatment with Renin-Angiotension System (RAS) blockers and SGLT-2 inhibitors for a minimum of 4 weeks prior to inclusion
* Safe contraception if women in childbearing age

Study B (patients with PKD):

* Prior diagnose with PKD
* eGFR >30 ml/min/1,73m2
* Treatment with Renin-Angiotension System (RAS) blockers for a minimum of 4 weeks prior to inclusion
* Safe contraception if women in childbearing age

Exclusion Criteria (Study A+B)

* Diabetes Mellitus type 1
* Heart Failure
* Liver Disease
* Kidney transplant
* Malignant diseases (except skin cancer)
* Recent acute myocardial infarction (AMI), apoplexia/transient ischemic attack (TIA) (within 3 months of inclusion)
* Pregnancy or breast feeding
* Alcohol or drug abuse
* Periodic fasting within four weeks of inclusion
* Routinely intake of ketogenic diet within four weeks of inclusion
* Treatment with nitrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proteinuria | Measured on 24 hour urine collection on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between Log UACR after 4 weeks treatment with ketone bodies and placebo (primary outcome study a)
GFR | Measured on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between GFR measured by Technetium99 (Tc99m) - Diethylene Triamine Pentaacetic Acid (DTPA) clearance after 4 weeks treatment with ketone bodies and placebo (primary outcome study b, secondary outcome in study a)

SECONDARY OUTCOMES:
Aldosterone | Measured on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference in plasma levels of aldosterone (pmol/L) after 4 weeks treatment with ketone bodies and placebo
P-Beta-hydroxybutyrate | Measured on the last day in each treatment period (each treatment period is 4 weeks)
  Change ind p-beta-hydroxybutyrate concentration
Excretion rate of renal tubular transport proteins | Measured on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between urine excretion rate of aquaporin 2 (AQP2) (pq/min), thiazide-sensitive sodium-chloride cotransporter (NCC)(pg/min), and distal epithelial sodium channel (ENaC)(pg/min) after 4 weeks treatment with ketone bodies and placebo
24-hour Ambulatory Blood Pressure | Measured using a Mobil-o-graph on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between systolic and diastolic 24-hour ambulatory blood pressure (mmHg) after treatment with ketone bodies and placebo.
Sodium and potassium excretion | Measured on 24 hour urine collection on the last day in each treatment period (each treatment period is 4 weeks)
  Diffeence between mean fractional and absolute excretion af sodium and postassium after 4 weeks treatment with ketone bodies and placebo
Peripherial Vascular Resistance | Measured using a Mobil-o-graph on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between peripherial vascular resistance (dyn*s/cm5) during treatment with ketone bodies compared to placebo
Heart rate | Measured using a Mobil-o-graph on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between heart rate after 4 weeks treatment with ketone bodies and placebo
Pulse Wave Velocity | Measured using a Mobil-o-graph on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference between pulse wave velocity (m/s) after 4 weeks treatment with ketone bodies and placebo
Renin | Measured on the last day in each treatment period (each treatment period is 4 weeks)
  Mean difference in plasma concentration of renin(pmol/L) after 4 weeks treatment with ketone bodies and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Trine Z Lyksholm, MD, Principal Investigator — University Clinic in Nephrology and Hypertenion, Godstrup Region Hospital
Locations (1):
- University Clinic in Nephrology and Hypertension, Gødstrup Region Hospital, Herning, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No